CLINICAL TRIAL: NCT00040638
Title: Phase 2 Study of TLK286 Administered Weekly in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, M.D. Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2014
Record Dates: First submitted 2002-07-02; First posted 2002-07-04 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TER 286

INTERVENTIONS:
Drug: TLK286

SUMMARY:
The purpose of this study is to determine the effectiveness of TLK286 in the treatment of advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non-small cell lung carcinoma
* Progressed while on or after treatment on platinum-based regimen
* Patients may not have had more than one prior cytotoxic chemotherapy regimen
* Stage IV or IIIB
* Age at least 18 years
* Adequate liver and kidney function
* Adequate bone marrow function

Exclusion Criteria:

* Pregnancy or lactation
* Unstable medical conditions
* Chemotherapy, hormonal therapy, radiotherapy, radiopharmaceuticals or immunotherapy within 3 weeks of TLK286
* CNS metastasis unless controlled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA Medical Center, Los Angeles, California
  - M.D. Anderson Cancer Center, Houston, Texas